CLINICAL TRIAL: NCT01470027
Title: N-Acetylcysteine for Neuroprotection in Parkinson's Disease
Acronym: NAC for PD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1109011912; 1R21AG041509 (NIH)
Record Dates: First submitted 2011-11-04; First posted 2011-11-10 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Parkinson Disease
Keywords: magnetic resonance spectroscopy; N-acetylcysteine; antioxidant; glutathione
MeSH Terms: conditions — Parkinson Disease | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- N-acetylcysteine 1800mg (Active Comparator): N-acetylcysteine 1800mg/day for 30 days
  Interventions: Drug: N-acetylcysteine
- N-acetylcysteine 3600mg (Active Comparator): N-acetylcysteine 3600mg daily for 30 days
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Placebo effervescent tablets daily for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — 900mg NAC effervescent tablets
  Other Names: NAC
  Arms: N-acetylcysteine 1800mg; N-acetylcysteine 3600mg
Drug: Placebo — effervescent tablets
  Arms: Placebo

SUMMARY:
The overall objective of this developmental/exploratory study is to use noninvasive proton magnetic resonance spectroscopy (1H MRS) to assess (a) whether brain levels of the antioxidant glutathione (GSH) are decreased in vivo, as has been found in postmortem brain, in 30 patients with Parkinson's disease (PD) compared to matched controls; (b) whether GSH levels in PD brain increase significantly following 30 days of daily supplementation with 1800mg or 3600mg of N-acetylcysteine (NAC) compared to placebo and to baseline, and (c) whether any such increases in brain GSH would be dose-dependent and be associated with a change in the participants' oxidative stress profiles. In addition, a clinical assessment battery, including quantitative tests of motor function, will be performed to investigate potential associations between the NAC intervention, brain GSH levels, oxidative stress markers, and clinical presentation. If successful, this study will represent the first objective documentation of whether there is a GSH deficit in living PD brain that dietary NAC supplementation can mitigate, thereby providing a compelling justification for investigating such neuroprotective strategies in larger controlled clinical trials.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder in which deficits of the primary intracellular antioxidant, glutathione (GSH), are postulated to mediate increased oxidative stress and mitochondrial dysfunction in the pathogenic cascade leading up to the loss of nigrostriatal dopaminergic neurons that is the hallmark of the disorder. Therefore, there is currently great interest in treatment strategies that can maintain, restore and/or elevate intracellular GSH levels. However, GSH does not readily cross the blood-brain barrier or the membranes of most cells, including neurons, so that direct dietary supplementation of the antioxidant has not proved viable in increasing its intracellular concentration. On the other hand, since the bioavailability of cysteine, which does cross both the blood-brain barrier and most cell membranes, is rate-limiting in the GSH synthesis pathway, this amino acid and its non-toxic derivatives, such as N-acetylcysteine (NAC), are being investigated as potential precursors that can be supplied through dietary means to spur in situ synthesis and elevation of brain GSH. The overall objective of this Exploratory/Developmental (R21) study is to use noninvasive proton magnetic resonance spectroscopy (1H MRS) to determine (a) whether levels of GSH are decreased in vivo in the brain of 30 patients with Parkinson's disease (PD) compared to matched controls, as has been found in postmortem brain; (b) whether GSH levels in PD brain increase significantly following 30 days of daily supplementation with 1800mg or 3600mg of NAC compared to baseline and placebo, and (c) whether any such increases in brain GSH would be dose-dependent and be associated with a change in the participants' oxidative stress profiles. Additionally, a clinical assessment battery, including quantitative tests of motor function, will be performed to investigate potential associations between the NAC intervention, brain GSH levels, oxidative stress markers, and clinical presentation. If successful, this study will represent the first objective documentation of whether there is a GSH deficit in living PD brain that dietary NAC supplementation can mitigate, thereby providing a compelling justification for investigating such neuroprotective strategies in larger controlled clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD according to the United Kingdom Parkinson's Disease Society Brain Bank criteria (UKPDSBB) criteria (only for PD group
* Age 50 to 75 years
* Able to give informed consent for study participation
* Not on any medication for PD (anticholinergic agents allowed)

Exclusion Criteria:

* Unable to give informed consent
* Unable to undergo a brain MRI
* PD duration ≥15 years
* Receiving dopamine receptor blocking agents, including typical neuroleptics, prochlorperazine, and metoclopramide
* Diagnosis of major depression or other axis I psychopathology
* Modified Mini-Mental Status Exam (MMSE) ≤ 24/30
* Diagnosis of chronic or persistent illnesses that could affect oxidative stress status, such as diabetes or congestive heart failure
* Significant concomitant medical disease limiting life expectancy to less than 12 months from study inclusion
* Diagnosis of primary mitochondrial disorder, epilepsy, stroke, multiple sclerosis or other neurodegenerative diseases such as Alzheimer's disease or ALS

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dikoma C. Shungu, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment for this pilot clinical study started in March 2012, as the end of the study in August 2016, 23 of 30 PD patients and 27 of 30 healthy volunteers (HV) subjects - a total 50- had participated in the study. All subjects enrolled at the Weill Cornell Parkinson's Disease and Movement Disorders Institute, led by the study neurologist.
Pre-assignment Details: A total of 50 subjects enrolled into the study (23 PD patients and 27 HV subjects). Only 21 patients with PD and 26 HV subjects underwent the baseline assessments. Two PD patients and 1 HV subject were excluded from the study before assignment to groups. All exclusion were unrelated to the study protocol.
Period: Overall Study
Arm/Group | N-acetylcysteine 1800mg | N-acetylcysteine 3600mg | Placebo
Started | 16 | 15 | 16
Completed | 15 | 14 | 15
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- N-acetylcysteine 1800mg - Parkinson's Patient: Parkinson's patient
  N-acetylcysteine 1800mg/day for 30 days
  N-acetylcysteine: 900mg NAC effervescent tablets
- N-acetylcysteine 3600mg -Parkinson's Patient: Parkinson's patient
  N-acetylcysteine 3600mg daily for 30 days
  N-acetylcysteine: 900mg NAC effervescent tablets
- Placebo -Parkinson's Patient: Parkinson's patient
  Placebo effervescent tablets daily for 30 days
  Placebo: effervescent tablets
- N-acetylcysteine 1800mg - Healthy Volunteer: Healthy Volunteer
  N-acetylcysteine 1800mg/day for 30 days
  N-acetylcysteine: 900mg NAC effervescent tablets
- N-acetylcysteine 3600mg -Healthy Volunteer: Healthy Volunteer
  N-acetylcysteine 3600mg daily for 30 days
  N-acetylcysteine: 900mg NAC effervescent tablets
- Placebo -Healthy Volunteer: Healthy Volunteer
  Placebo effervescent tablets daily for 30 days
  Placebo: effervescent tablets
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer | Total
Number analyzed (Participants) | 7 | 7 | 7 | 9 | 8 | 9 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.000 (5.259) | 61.714 (6.264) | 62.429 (2.820) | 64.222 (7.807) | 56.625 (5.927) | 59.778 (5.995) | 60.809 (6.173)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 3 | 1 | 1 | 10
  Male | 6 | 6 | 4 | 6 | 7 | 8 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2 | 2 | 1 | 7
  Not Hispanic or Latino | 6 | 6 | 7 | 7 | 6 | 8 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 4 | 3 | 4 | 11
  White | 5 | 7 | 6 | 5 | 5 | 5 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 7 | 9 | 8 | 9 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change of Cerebral Glutathione Levels as Measured by Proton Magnetic Resonance Spectroscopy
Description: In vivo brain GSH measured with 1H MRS in the unmedicated patients with idiopathic PD and in sex- and age-matched healthy controls prior to and following 4 weeks supplementation with either placebo, 1800mg/day or 3600 mg/day of NAC. Striatal and occipital cortex glutathione levels as measured in vivo by 1H MRS at baseline and following 4 weeks of treatment with placebo, 1800mg NAC/day and 3600mg NAC/day.
  The area under the GSH spectral peak was obtained by frequency-domain fitting of the GSH resonance in the edited spectrum to a pseudo-Voigt lineshape function using a robust and highly optimized public-domain Levenberg-Marquardt nonlinear least-squares minimization routine. The resulting peak areas were then expressed as ratios relative to the synchronously acquired and similarly fitted unsuppressed voxel water signal.
Time Frame: at baseline and 4 weeks after intervention start
Population: The number of participants in the Participant Flow module is different from the Overall Number of Participants for brain GSH levels because of the total sample of 47 subjects enrolled in the study, baseline and post-treatment GSH values were available only for 43 subjects, whose data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer
Number analyzed (Participants) | 6 | 7 | 7 | 8 | 6 | 9
Ratio
  Baseline ( In Striatum) | 3.422 (0.7371) | 3.334 (0.8754) | 3.745 (1.418) | 4.282 (0.946) | 4.415 (0.928) | 3.901 (0.9698)
  4 weeks after intervention start ( In Striatum) | 3.404 (0.7684) | 3.473 (1.010) | 4.105 (1.292) | 4.843 (0.9884) | 3.900 (0.724) | 3.831 (0.8106)
  Baseline ( In Occipital) | 1.743 (0.4867) | 1.938 (0.3415) | 1.799 (0.4608) | 2.190 (0.5077) | 2.007 (0.395) | 2.001 (0.4755)
  4 weeks after intervention start ( In Occipital) | 1.962 (0.5012) | 2.108 (0.3788) | 2.118 (0.422) | 2.161 (0.4027) | 1.990 (0.3344) | 2.298 (0.7663)

2. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Parts I-V (Total Score Reported)
Description: The UPDRS is considered the gold standard for determining disease severity and progression in patients with Parkinson's disease. It consists of the following five elements:
  1. Evaluation of mentation, behavior and mood.
  2. Self evaluation of the activities of daily living (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, etc.
  3. Motor evaluation by a clinician.
  4. Hoehn and Yahr scale (Hoehn 1967) for the description of the overall disease severity in PD with 8 stages.
  5. Schwab and England activities of daily living scale (Schwab and England 1969) for the estimation of the general abilities in PD patients. The Schwab and England ADL scale is graduated in 10% steps with 100% indicating complete independence and 0% indicating an individual in whom the vegetative functions are completely impaired.
  A total of 199 points are possible for UPDRS, with 199 representing the worst disability and 0 no disability.
Time Frame: at baseline and 4 weeks after intervention start
Population: The number of participants in the Participant Flow module is different from the Overall Number of Participants for Unified Parkinson's Disease Rating Scale (UPDRS) because of the total sample of 47 subjects enrolled in the study, baseline and post-treatment UPDRS were available only for 40 subjects, whose data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 4 | 7
units on a scale
  Baseline | 35.286 (15.152) | 31.500 (10.782) | 16.714 (4.923) | 1.000 (2.071) | 4.500 (2.082) | 3.143 (5.429)
  4 weeks after intervention start | 23.857 (16.547) | 24.249 (16.547) | 13.857 (6.817) | 0.600 (1.342) | 3.000 (2.160) | 1.857 (3.185)

3. Secondary Outcome: Mini Mental State Examination (MMSE)
Description: The MMSE is a brief questionnaire-based test that is used to screen for cognitive impairment. Domains tested are orientation to time and place, registration, attention and calculation, recall, language, repetition and complex commands. Scores lower than 25/30 points indicate mild (21-24 points), moderate (10-20 points) or severe (<10 points) cognitive impairment, but scores may need to be corrected for educational attainment, age and interfering impairments such as motor deficits that affect drawing skills.
Time Frame: at baseline and 4 weeks after intervention start
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer
Number analyzed (Participants) | 7 | 7 | 7 | 9 | 8 | 9
units on a scale
  Baseline | 29.571 (0.5345) | 29.857 (0.3780) | 29.571 (0.787) | 29.778 (0.667) | 29.625 (0.518) | 30.000 (0.000)
  4 weeks after intervention start | 29.667 (0.516) | 29.714 (0.489) | 30.000 (0.000) | 29.857 (0.378) | 30.000 (0.000) | 29.750 (0.463)

4. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: The Hamilton Depression Rating Scale (HAM-D) is a 21-item instrument designed to measure the severity of illness in adults already diagnosed as having depression. The Hamilton Depression Rating Scale (HAM-D) has proven useful for many years as a way of determining a patient's level of depression before, during, and after treatment. It is clinician-administered and requires 15 to 20 minutes complete the interview and score the results. Although the HAM-D form lists 21 items, the scoring is based on the first 17. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2.
  The minimum score is 0 and maximum score is 50. The scale has been widely used in clinical practice and become a standard in pharmaceutical trials.
  HAM-D Scoring Instructions are following:
  0-7 = Normal; 8-13 = Mild Depression; 14-18 = Moderate Depression; 19-22 = Severe Depression;
  ≥ 23 = Very Severe Depression.
Time Frame: at baseline and 4 weeks after intervention start
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer
Number analyzed (Participants) | 7 | 7 | 7 | 9 | 8 | 9
units on a scale
  Baseline | 3.714 (2.430) | 3.571 (2.430) | 1.857 (1.951) | 2.222 (3.032) | 1.875 (1.807) | 1.889 (2.2608)
  4 weeks after intervention start | 4.167 (3.869) | 3.857 (2.854) | 1.714 (1.976) | 1.286 (1.890) | 0.714 (1.113) | 1.222 (1.922)

5. Secondary Outcome: 9-Hole Peg Board Test (9-HPT)
Description: The 9-HPT is a standardized, quantitative timed test of upper extremity motor function. Individuals are asked to place and remove nine pegs, one at a time, from nine holes in a board as quickly as possible. The task is performed twice with the dominant and twice with the non-dominant hand, and the average time to complete the task once is calculated for each hand. The 9-HPT has a high inter- and intra-rater reliability, is validated and is sensitive to detect minor impairments of hand function.
Time Frame: at baseline and 4 weeks after intervention start
Population: The measurement used for the 9-HPT is the average of time needed to complete the task with the dominant and non-dominant hand recorded in seconds. The presence of PD is expected to produce higher test times in seconds.
Measure: Mean (Standard Deviation); unit: s (in seconds)
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer
Number analyzed (Participants) | 7 | 7 | 7 | 9 | 8 | 9
s (in seconds)
  Baseline | 37.026 (19.509) | 27.795 (5.660) | 28.694 (7.886) | 25.088 (4.489) | 24.593 (6.089) | 25.834 (4.964)
  4 weeks after intervention start | 32.756 (7.116) | 25.980 (6.231) | 28.084 (9.373) | 24.940 (2.995) | 22.511 (6.325) | 24.704 (4.566)

6. Secondary Outcome: 10-Meter Walk Test
Description: The 10-meter walk test is a standardized, quantitative timed test of lower body motor function. The maximal gait speed is measured during a 10-meter walk. The task will be performed three times and the average time to complete the task once will be recorded. The 10-meter walk test is a reliable and sensitive measure of gait function in elderly individuals and PD patients.
  Cut-off values:
  < 0.4 m/s more likely to be household ambulators; 0.4 - 0.8 m/s limited community ambulators; > 0.8 m/s community ambulators.
Time Frame: at baseline and 4 weeks after intervention start
Population: The number of participants in the Participant Flow module is different from the Overall Number of Participants for 10-Meter Walk Test because of the total sample of 47 subjects enrolled in the study, baseline and post-treatment 10-Meter Walk Test score were available only for 46 subjects, whose data were included in the analysis.
Measure: Mean (Standard Deviation); unit: m/s (meters per second)
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer
Number analyzed (Participants) | 7 | 7 | 7 | 9 | 8 | 8
m/s (meters per second)
  Baseline | 7.816 (1.820) | 7.289 (1.281) | 6.896 (0.907) | 7.253 (0.713) | 10.403 (6.380) | 7.141 (0.929)
  4 weeks after intervention start | 10.513 (7.136) | 7.434 (1.389) | 6.296 (0.929) | 7.279 (0.643) | 9.740 (5.958) | 6.893 (0.937)

7. Secondary Outcome: Beck Anxiety Inventory
Description: The Beck Anxiety Inventory (BAI) is a clinician-administered and validated instrument to discriminate anxiety from depression. The standardized BAI cutoffs are:
  0-9: minimal anxiety; 10-16: mild anxiety; 17-29: moderate anxiety; 30-63: severe anxiety.
Time Frame: at baseline and 4 weeks after intervention start
Population: The number of participants in the Participant Flow module is different from the Overall Number of Participants for Beck Anxiety Inventory (BAI) test because of the total sample of 47 subjects enrolled in the study, baseline and post-treatment BAI scores were available only for 45 subjects, whose data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer
Number analyzed (Participants) | 6 | 7 | 7 | 9 | 8 | 8
units on a scale
  Baseline | 7.000 (6.782) | 9.000 (5.686) | 6.333 (5.046) | 3.778 (4.944) | 3.750 (5.365) | 2.625 (3.067)
  4 weeks after intervention start | 3.000 (2.450) | 8.286 (4.386) | 5.714 (5.438) | 2.429 (2.371) | 5.714 (5.345) | 4.333 (8.789)

8. Secondary Outcome: Parkinson's Disease Quality of Life Questionnaire (PDQLQ)
Description: The Parkinson's Disease Quality of Life Questionnaire is a self completion PRO designed to address aspects of functioning and well-being for those affected by Parkinson's disease.
  The Parkinson's Disease Quality of Life Questionnaire is coded on a scale of 0 to 185, with 185 indicating perfect health and 0 indicating very poor health.
Time Frame: at baseline and 4 weeks after intervention start
Population: The number of participants in the Participant Flow module is different from the Overall Number of Participants for PDQLQ because of the total sample of 47 subjects enrolled in the study, baseline and post-treatment PDQLQ scores were available only for 43 subjects, whose data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer
Number analyzed (Participants) | 6 | 7 | 6 | 9 | 8 | 8
units on a scale
  Baseline | 134.333 (34.488) | 142.285 (14.739) | 159.833 (13.586) | 175.667 (19.526) | 171.625 (18.647) | 175.250 (14.008)
  4 weeks after intervention start | 127.100 (45.081) | 135.571 (14.010) | 159.429 (17.634) | 177.833 (11.565) | 165.142 (17.601) | 181.750 (2.964)

ADVERSE EVENTS:
Time Frame: Baseline (day 0) to 4 weeks after intervention start
Arm/Group | N-acetylcysteine 1800mg - Parkinson's Patient | N-acetylcysteine 3600mg -Parkinson's Patient | Placebo -Parkinson's Patient | N-acetylcysteine 1800mg - Healthy Volunteer | N-acetylcysteine 3600mg -Healthy Volunteer | Placebo -Healthy Volunteer
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/9 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/9 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 2/7 | 2/7 | 2/7 | 2/9 | 2/8 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine 1800mg - Parkinson's Patient (N=7) | N-acetylcysteine 3600mg -Parkinson's Patient (N=7) | Placebo -Parkinson's Patient (N=7) | N-acetylcysteine 1800mg - Healthy Volunteer (N=9) | N-acetylcysteine 3600mg -Healthy Volunteer (N=8) | Placebo -Healthy Volunteer (N=9)
nausea and vomiting, loss of appetite (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Few days of nausea and vomiting, loss of appetite, no stomach pain
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) — Headache, neck pain, tiredness
Incidental finding in MRI (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — left Acom aneurysm - intervention unwarranted due to small size
Shoulder and neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Doctor think it is due to a rotatory cuff
Occasional skin itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Occasional skin itching
Metallic taste, Occasional light-headed on standing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
puffy face, increased heart rate (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Withdrew from study. Described "hot flash inside head"
Lightheaded after exercise, daytime napping (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was limited by recruitment challenges related to identifying sufficient numbers of patients with PD who met all the eligibility criteria, especially with respect to medication status, and were willing to enter into the 4-week trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No